CLINICAL TRIAL: NCT06054984
Title: To Investigate the Safety, Tolerability, Efficacy and Pharmacokinetics of T Cell Receptor T Cell Therapy in the Treatment of Advanced Pancreatic Cancer
Brief Title: TCR-T Cells in the Treatment of Advanced Pancreatic Cancer
Acronym: GB3010-02
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: Shanghai Essight Bio Co.,Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: (2021) IEC No.288
Record Dates: First submitted 2023-03-31; First posted 2023-09-26 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-03

CONDITIONS: Pancreatic Cancer
Keywords: TCR-T; T cells; RAS; TP53; Cell therapy
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients were sequentially enrolled into 3 dose escalation groups(dose level 1 to 3):5×10^8±20%,5×10^9±20%,5×10^10±20%. Twenty-eight days after infusion of GB3010 cells was the observation period for DLT evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCR-T Cells Injection（GB3010 Cells Injection） (Experimental): This study was designed to evaluate the safety, tolerability, efficacy, and pharmacokinetics of TCRT cell injection (GB3010) in patients with advanced pancreatic cancer by intravenous injection. The target population is patients with advanced pancreatic cancer who lack effective treatment methods, so that the benefits of patients participating in clinical trials will outweigh the risks.
  Interventions: Drug: TCR-T Cells Injection（GB3010 Cells Injection）

INTERVENTIONS:
Drug: TCR-T Cells Injection（GB3010 Cells Injection） — The TCRT cells used in this clinical trial were derived from the patient's autologous peripheral-blood T cells and were genetically transduced to express a T-cell Receptor that recognizes the RAS/TP53.Patients were sequentially enrolled into 3 dose escalation groups(dose level 1-3) :5×10^8±20%,5×10^9±20%,5×10^10±20%.

SUMMARY:
To investigate the safety, tolerability, efficacy and pharmacokinetics of TCR-T cells in the treatment of advanced pancreatic cancer

DETAILED DESCRIPTION:
The aim of this clinical trial is to investigate the safety, tolerability, efficacy and pharmacokinetics of TCR-T cell therapy in patients with advanced pancreatic cancer by intravenous injection, in order to explore an effective cellular immunotherapy method for the treatment of advanced pancreatic cancer

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for the study, patients must meet all of the following criteria:

  1. Male or female, aged 18-75 years;
  2. Patients with advanced pancreatic cancer diagnosed by histology or cytology, patients who failed to respond to standard treatment, relapsed or voluntarily gave up;
  3. Patients must have tumor tissue that expresses specific tumor antigens, such as mutations in RAS and/or TP53;
  4. Patients must undergo HLA matching testing and meet the requirements of HLA matching.
  5. At least one measurable or evaluable lesion ≥15 mm according to RECIST1.1 criteria;
  6. Patients with ECOG < 2 and life expectancy ≥3 months;
  7. a) Liver function: ALT/AST < 3 times the upper limit of normal value (ULN) and bilirubin ≤34.2μmol/L; b) renal function: creatinine < 220μmol/L; c) terminal oxygen saturation ≥95% in room air; d) Cardiac function: left ventricular ejection fraction (LVEF) ≥60%; e) Blood routine: absolute neutrophil count ≥ 1×109/L; Platelet count ≥70×109/L; Absolute lymphocyte count ≥100 cells /μL;
  8. The patients met the requirements of apheresis without any contraindications.
  9. Women of childbearing age who have a negative urine pregnancy test at screening and before starting dosing and who have agreed to use highly effective contraception for at least 100 days after infusion; Female participants must agree not to donate eggs (oocytes, oocytes) for assisted reproductive purposes during the study and for 90 days after receiving the last study drug;
  10. Male subjects with a fertile partner must consent to use an effective barrier method of contraception for at least 100 days after infusion; Must agree not to donate sperm for at least one year;
  11. Sign an informed consent form.

Exclusion Criteria:

* Patients who met any of the following criteria were not eligible for inclusion in the study:

  1. Persons with severe mental disorders;
  2. A positive virological test for any of the following: HIV; HCV; HBsAg; HBcAb was positive, and HBV DNA copy number and TPPA were positive.
  3. Patients with severe allergic history or allergic constitution;
  4. Severe underlying medical conditions such as evidence of other serious active viral, bacterial or uncontrolled systemic fungal infection; Active autoimmune disease or a history of autoimmune disease within 3 years;
  5. A history of autoimmune diseases (e.g., Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus) leading to end-organ damage or requiring systemic immunosuppressive/systemic disease modulating drugs within the past 2 years;
  6. Combined with organ dysfunction, such as renal insufficiency;
  7. Had been enrolled in another clinical trial within 4 weeks before enrollment in the trial;
  8. Those who were unable to comply with the study protocol and follow-up plan due to physiological, family, social, geographical and other factors;
  9. Patients with contraindications to cyclophosphamide or fludarabine chemotherapy;
  10. Subjects who required additional immunosuppressive drug therapy within 72 hours before TCR-T infusion, except for the treatment of adverse events during the trial;
  11. Pregnant, lactating women, or men who plan to have children while participating in the study or within 100 days of receiving study treatment;
  12. Any other condition considered by the investigator to be ineligible for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-09-07 (Actual); Primary Completion 2024-06-07 (Estimated); Study Completion 2024-09-07 (Estimated)

PRIMARY OUTCOMES:
Evaluate the Incidence of Treatment Related Adverse Events of TCRT cells in patients with advanced pancreatic cancer | 2years
  collect adverse events (AE), serious adverse events (SAE), adverse events of special interest (AESI), and laboratory abnormalities (type, frequency, and severity)
Characterize the Peak of Peripheral Blood Concentration and Area under the Peripheral Blood concentration versus time curve of TCRT cells and observe their proliferation and persistence in body | 2years
  After infusion of neoantigen-specific TCRT cells, collect peak (Cmax) of neoantigen-specific TCRT cells in blood and tumor tissue, time to peak (number of days to peakTCRT cells after infusion), Tmax) and AUC0-28 (area under the curve plotted against visit time by the number of neoantigen-specific TCRT cells in peripheral blood from day 0 to 28). "If possible, AUC0-inf, terminal phase elimination rate constant (λz), elimination half-life (t1/2) will be evaluated."

SECONDARY OUTCOMES:
Correlation of the pharmacokinetic profile of TCRT cells with the Incidence of CRS and ICANS events | 2years
  collect changes in mutant cell concentration in peripheral blood and tumor tissue after TCRT cell reinfusion,observe correlation of these measures with CRS and ICANS events
Evaluate tumor size (mm) , tumor biomarker CA19-9 (U/ml), ORR/DCR/PFS and OS of patients with advanced pancreatic cancer | 2years
  ORR at 2, 4, and 6 months after TCRT cell infusion (ORR=CR+PR). The primary efficacy outcome was the change in target tumor size (local control rate of target lesions). Secondary efficacy indicators: changes in tumor markers; Objective response rate (ORR), disease control rate (DCR), progression-free survival (PFS) and overall survival (OS) according to RECIST1.1 criteria

OTHER OUTCOMES:
To explore the correlation between the proliferation and persistence of TCRT cells in body and the efficacy | 2years
  observe correlation of the PK parameters with response (CR, PR, relapse),PK parameters including peak (Cmax) of neoantigen-specific TCRT cells in blood and tumor tissue, time to peak (number of days to peakTCRT cells after infusion), Tmax) and AUC0-28 (area under the curve plotted against visit time by the number of neoantigen-specific TCRT cells in peripheral blood from day 0 to 28).

CONTACTS AND LOCATIONS:
Overall Officials: BoYongShen, Study Director — Ruijin Hospital
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China